CLINICAL TRIAL: NCT03548675
Title: Pharmacogenetics to Improve Personalized Antidepressant Dosing in Patients With Severe Depression;a Randomized Controlled Trial Using Tricyclic Antidepressants
Brief Title: Pharmacogenetics Informed Tricyclic Antidepressant Dosing (PITA)
Acronym: PITA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 848016004
Record Dates: First submitted 2018-05-23; First posted 2018-06-07 (Actual); Last update posted 2022-11-29 (Actual); Status verified 2022-11

CONDITIONS: Depressive Disorder, Major
Keywords: Pharmacogenetics; Antidepressive Agents
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Intervention Model Description: This study is a randomized controlled clinical trial.
Who Masked: Outcomes Assessor
Masking Description: Prescribing physicians will be unblinded for the genotype and the resulting metabolization phenotype. Outcome assessments will be performed by blinded researchers and the patients themselves (self-assessments).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Genotype-guided TCA treatment (Experimental): Genotype guided dosing of the TCAs in patients with a PM,IM,EM or UM phenotype based on pharmacogenetic test.
  Interventions: Drug: TCA treatment
- Standard TCA treatment (Active Comparator): Standard dosing of TCA in patients with a PM,IM, EM or UM phenotype based on pharmacogenetic test
  Interventions: Drug: TCA treatment

INTERVENTIONS:
Drug: TCA treatment — All patients fulfilling inclusion criteria will be genotyped for CYP2C19 and CYP2D6 genes. Based on the genetic test results patients will be classified into a metabolisation phenotype (UM, EM, IM or PM).

SUMMARY:
Tricyclic Antidepressants (TCA's) are the cornerstone of treatment for patients with severe Major Depressive Disorder (sMDD). Current dosing is guided by repeated measurements of blood levels. Compared to patients with a normal metabolization function, for those with increased CYP450 enzyme activity it takes longer to reach a therapeutic drug level. The consequent delay of drug efficacy is associated with a prolonged treatment period, increased risk of suicidal behaviour and eventually lower remission rates. For those with reduced CYP450 activity higher rates of side effects are expected. An innovative TCA dosing strategy, taking the genetic variants of CYP2D6 and CYP2C19 into account may help to reduce the above mentioned problems. Up till now, the current guidelines for CYP450 pharmacogenetics based TCA dosing have not been systematically evaluated for effectiveness and cost-effectiveness in larger groups of patients. Such evaluation is necessary before broad implementation of these guidelines can be advocated. In the present study 200 patients with sMDD who are treated with nortriptyline, clomipramine or imipramine are randomized over two strategies: dosing based both on CYP450-genotype and blood level measurements and dosing as usual (standard doses plus blood levels). We hypothesize that genotype informed dosing results in faster attainment of therapeutic drug levels, lower rates of side effects, earlier symptom relief and lower levels of health- and working related costs.

ELIGIBILITY:
Inclusion Criteria:

Patients are in- and outpatients, having a primary diagnosis of severe major depressive disorder (SCID-I diagnosis in agreement with DSM-5 criteria and a Hamilton Rating Scale for Depression score ≥ 19 (HAM-D-17-item version), aged 18-65 years, who, according to their physician, are eligible for treatment with a TCA (Nortriptyline (NOR), Clomipramine (CLOMI) or Imipramine (IMI)). The choice of the specific TCA is at the discretion of the physician in attendance.

Exclusion Criteria:

1. Psychotic depression
2. Bipolar I or II disorder.
3. Schizophrenia or other primary psychotic disorder.
4. Drug or alcohol dependence in the past 3 months.
5. Mental Retardation (IQ < 80).
6. For women: pregnancy or possibility for pregnancy without adequate contraceptive measures.
7. Breastfeeding.
8. Serious medical illness affecting the CNS, including but not restricted to M Parkinson, SLE, brain tumour, CVA.
9. Relevant medical illness as contra-indication for TCA use, such as recent myocardial infarction.
10. Other drugs influencing the pharmacokinetics of the TCAs as based on a list of interacting drugs. In case of psychotropic co-medication only a benzodiazepine in a dose equivalent up to 4 mg lorazepam will be allowed.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2018-05-23 (Actual); Primary Completion 2022-02-02 (Actual); Study Completion 2022-07-13 (Actual)

PRIMARY OUTCOMES:
Time to TCA plasma concentration in the therapeutic range | During the 7 weeks treatment phase
  Time to TCA plasma concentration in the therapeutic range

SECONDARY OUTCOMES:
Reduction of depressive symptoms | Difference between measurements at baseline and after 7 weeks of treatment
  HAM-D reduction
Highest level of side effects | During the 7 weeks treatment phase
  summary measure: FIBSER
Economic Evaluation (Cost Effectiveness) | 26 weeks after the start of treatment
  Utility based on EQ5D5L measurement

CONTACTS AND LOCATIONS:
Overall Officials: Joost Janzing, MD PhD, Principal Investigator — Radboudumc dept of Psychiatry
Locations (1):
- Radboudumc Dept of Psychiatry, Nijmegen, Netherlands

REFERENCES:
- [Derived] Dalhuisen I, Biemans T, Vos CF, Hark ST, van Oostrom I, Spijker J, Wijnen B, van Exel E, van Mierlo H, de Waardt D, Arns M, Tendolkar I, Janzing J, van Eijndhoven P. A comparison between rTMS and antidepressant medication on depressive symptom clusters in treatment-resistant depression. Eur Arch Psychiatry Clin Neurosci. 2025 Sep;275(6):1799-1807. doi: 10.1007/s00406-025-02012-0. Epub 2025 Apr 23. PMID 40266345
- [Derived] Vos CF, Ter Hark SE, Schellekens AFA, Spijker J, van der Meij A, Grotenhuis AJ, Mihaescu R, Kievit W, Donders R, Aarnoutse RE, Coenen MJH, Janzing JGE. Effectiveness of Genotype-Specific Tricyclic Antidepressant Dosing in Patients With Major Depressive Disorder: A Randomized Clinical Trial. JAMA Netw Open. 2023 May 1;6(5):e2312443. doi: 10.1001/jamanetworkopen.2023.12443. PMID 37155164